CLINICAL TRIAL: NCT00943085
Title: Family-Focused Therapy as Early Treatment for Youth at Risk for Bipolar Disorder
Brief Title: Early Family-Focused Treatment for Youth at Risk for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH077856 (NIH); R34MH077856 (NIH); 5R34MH077856 (NIH); DSIR 84-CTS
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Disorder
Keywords: Early Signs of Bipolar Disorder; High Risk Youth; Adolescence; Childhood
MeSH Terms: conditions — Bipolar Disorder | interventions — Family Therapy; Psychosocial Intervention; Psychotherapy; Behavior Therapy; Crew Resource Management, Healthcare; Diagnostic Self Evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-focused therapy (Experimental): Participants will receive family-focused therapy.
  Interventions: Behavioral: Family-focused therapy
- Brief educational treatment (Active Comparator): Participants will receive one session of diagnostic feedback, recommendations for continued treatment, and crisis intervention as needed.
  Interventions: Behavioral: Brief educational treatment

INTERVENTIONS:
Behavioral: Family-focused therapy — 12 therapy sessions involving the at-risk child or adolescent, parents, and available siblings. Therapy will include psychoeducation about mood disorders, communication enhancement training, and problem-solving skills training. Ongoing medication management from a study psychiatrist will be available.
  Other Names: FFT; Family Therapy; Psychoeducation; Psychosocial Intervention; Psychotherapy; Behavior Therapy
  Arms: Family-focused therapy
Behavioral: Brief educational treatment — Thorough diagnostic assessment by a study evaluator, separate evaluation by a child psychiatrist, feedback session with parents and child, and provision of reading materials pertinent to managing childhood mood disorders. Ongoing medication management and crisis-oriented family sessions will be available as needed.
  Other Names: Psychoeducation; Crisis Management; Enhanced Care; Diagnostic Evaluation
  Arms: Brief educational treatment

SUMMARY:
This study will test a family-based therapy aimed at preventing or reducing the symptoms of bipolar disorder in at-risk children.

DETAILED DESCRIPTION:
Early-onset bipolar disorder (BD) is a chronic, recurrent disorder that starts before age 18. In addition to the debilitating effects of BD, which include episodes of lethargic depression and exhausting mania, children and adolescents with BD often have co-occurring disorders, such as attention deficit hyperactivity disorder, conduct disorder, substance abuse disorders, and anxiety disorders. Early interventions may lead to better mental health by preventing BD from ever fully expressing itself. This study will test an early intervention for BD called family-focused treatment (FFT), which targets children and adolescents who are at risk for developing BD. FFT will include education about BD and training in communication strategies and problem-solving skills. It will focus on the family, because family environmental factors are related to the course and recurrence of BD. By reducing risk factors and teaching coping skills, FFT aims to prevent expression of BD, delay the onset or reduce the severity of manic episodes, and ensure that the first treatment received is appropriate.

Participation in this study will last 1 year and include three parts. In the first part, participating children and their families will complete research interviews and questionnaires about the child's mood, behavior, beliefs, and problems. Parent participants will also provide information on the family background of mood or anxiety problems. In the second part, participants will be randomly assigned to receive one of two treatments: FFT or brief educational treatment. Participants receiving FFT will complete 12 therapy sessions in which parents, children, and siblings learn how to cope with mood disorders, new ways to talk to each other, and strategies for solving family problems. FFT sessions will occur weekly for the first 8 weeks and then every other week for the next 8 weeks. Participants receiving brief educational treatment will complete diagnostic assessments and a 1-hour individualized feedback session, and they will be given a workbook about childhood mood disorders. A counselor will be available to all participants, in case of emergencies, for the full study year. All participants will also be provided with standard pharmacotherapy as needed. In the third part of the study, participants will complete follow-up assessments every 4 months for 1 year. Assessments will include interviews and questionnaires similar to those completed in the first part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one biological parent or stepparent with whom the child or adolescent participant lives and who is willing to participate in family treatment
* Has a DSM-IV diagnosis of at least one of the following within the past 2 years : bipolar disorder not otherwise specified (BD-NOS), major depressive disorder (MDD), or cyclothymia
* If the main diagnosis is MDD, the depressive episode must have occurred within the past 2 years
* Has evidence of current significant affective symptoms, as determined by a score greater than 11 on the Young Mania Rating Scale within the last week or a score greater than 29 on the Child Depression Rating Scale-Revised within the last 2 weeks
* Not currently enrolled in family or marital therapy
* Has at least one biological parent or sibling with a verifiable diagnosis of bipolar disorder I or II
* Speaks English

Exclusion Criteria:

* Fully diagnosable bipolar disorder I or II
* Diagnosis of autism or pervasive developmental disorder
* Evidence of mental retardation, as defined by an intelligence quotient (IQ) less than 70
* Presence of comorbid neurologic diseases such as seizure disorder
* Substance or alcohol abuse or dependence disorders in the 4 months prior to study recruitment
* Evidence of a life-threatening eating disorder or other medical disorder that requires emergency medical treatment
* Has previously been treated with family-focused therapy
* Evidence of current sexual or physical abuse or domestic abuse between the adult partners

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in symptoms and functioning of at-risk children, as defined by depression and mania scores and psychiatric status on the Adolescent Longitudinal Interval Follow-up Evaluation (A-LIFE) | Measured every 4 months for 1 year

SECONDARY OUTCOMES:
Delayed onset of first manic, mixed, or hypomanic episode, measured on the A-LIFE | Measured every 4 months for 1 year
Scores on the Child Depression Rating Scale | Measured every 4 months for 1 year
Scores on the Young Mania Rating Scale | Measured every 4 months for 1 year
Parental mood and distress, as measured by the Beck Depression Inventory, Symptom Checklist | Measured every 4 months for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David J. Miklowitz, PhD, Principal Investigator — University of Colorado, Boulder
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Lucile Packard Children's Hospital, Stanford, California
  - University of Colorado, Boulder, Boulder, Colorado

REFERENCES:
- [Background] Miklowitz DJ, Chang KD. Prevention of bipolar disorder in at-risk children: theoretical assumptions and empirical foundations. Dev Psychopathol. 2008 Summer;20(3):881-97. doi: 10.1017/S0954579408000424. PMID 18606036
- [Background] Chang K, Howe M, Gallelli K, Miklowitz D. Prevention of pediatric bipolar disorder: integration of neurobiological and psychosocial processes. Ann N Y Acad Sci. 2006 Dec;1094:235-47. doi: 10.1196/annals.1376.026. PMID 17347355
- [Result] Miklowitz DJ, Schneck CD, Singh MK, Taylor DO, George EL, Cosgrove VE, Howe ME, Dickinson LM, Garber J, Chang KD. Early intervention for symptomatic youth at risk for bipolar disorder: a randomized trial of family-focused therapy. J Am Acad Child Adolesc Psychiatry. 2013 Feb;52(2):121-31. doi: 10.1016/j.jaac.2012.10.007. Epub 2013 Jan 2. PMID 23357439
- [Derived] Schneck CD, Chang KD, Singh MK, DelBello MP, Miklowitz DJ. A Pharmacologic Algorithm for Youth Who Are at High Risk for Bipolar Disorder. J Child Adolesc Psychopharmacol. 2017 Nov;27(9):796-805. doi: 10.1089/cap.2017.0035. Epub 2017 Jul 21. PMID 28731778
- See also: UCLA Child and Adolescent Mood Disorders Program — http://www.semel.ucla.edu/champ